CLINICAL TRIAL: NCT04742985
Title: Effects of Combined Extracts of Green Tea Seed (Saponins) and Green Tea Leaves (Epigallocatechin-3-gallate) on Gastric Mucosal Protection: A Pilot Study
Brief Title: Effects of Green Tea Extracts on Gastric Mucosal Protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2020-048
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Green tea combined extracts group A (Experimental): This group takes Green tea combined extracts (62.5 mg) for 8 weeks.
  Interventions: Dietary Supplement: Green tea combined extracts group
- Green tea combined extracts group B (Experimental): This group takes Green tea combined extracts (125 mg) for 8 weeks.
  Interventions: Dietary Supplement: Green tea combined extracts group
- Placebo group (Placebo Comparator): This group takes placebo for 8 weeks.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Green tea combined extracts group — Green tea combined extracts 320 mg/day (main compound 62,5 mg for A group, 125 mg for B group) during 8 weeks
  Arms: Green tea combined extracts group A; Green tea combined extracts group B
Dietary Supplement: Placebo group — Placebo 320 mg/day during 8 weeks
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled pilot study to investigate the effects of a combined extract of green tea seed (saponins) and green tea leaves (epigallocatechin-3-gallate) on gastric mucosal protection in adults with functional dyspepsia for 8 weeks.

DETAILED DESCRIPTION:
A previous study has indicated that combined extract of green tea seed (saponins) and green tea leaves (epigallocatechin-3-gallate) may improve gastric mucosal status in rat with alcohol-induced gastritis.Therefore, the investigators conduct a randomized, double-blind, placebo-controlled pilot study to investigate the effects of a combined extract of green tea seed (saponins) and green tea leaves (epigallocatechin-3-gallate) on gastric mucosal protection in adults with functional dyspepsia for 8 weeks; the safety of the compound are also evaluated. The Investigators examine C-reactive protein, IFN-γ, TNF-α, gastrin, malondialdehyde, 8-hydroxy-2' -deoxyguanosine, and questionnaires (Gastrointestinal Symptom Rating Scale, Nepean dyspepsia index-Korean version, Nepean dyspepsia index-Korean version QOL questionnaire, Gastrointestinal symptom scale) at baseline and after 8 weeks of intervention. Twenty four adults were administered either 320 mg of combined extracts of green tea seed (saponins) and green tea leaves (epigallocatechin-3-gallate) or a placebo each day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The Rome IV criteria define dyspepsia as any combination of 4 symptoms: postprandial fullness, early satiety, epigastric pain, and epigastric burning that are severe enough to interfere with the usual activities and occur at least 3 days per week over the last 3 months

Exclusion Criteria:

* Patients complaining of severe gastrointestinal symptoms requiring immediate medication
* Those with a history of gastric acid hypersecretion such as Zollinger-Ellison Syndrome
* Those who received Helicobacter pylori eradication therapy within 4 weeks
* Those who have taken nonsteroidal anti-inflammatory drugs, steroid drugs or antibiotics, aspirin or antithrombotic drugs, or gastric acid suppressants within 4 weeks
* Those who have a history of upper gastrointestinal tract surgery, stenosis, bleeding, esophageal dilatation, gastric mucosal resection, etc. within the past 1 year
* Patients with gastric ulcer (active or healing), duodenal ulcer (active or healing), reflux esophagitis (LA B or higher), or malignant tumors from gastroscopy performed within the last 6 months
* Abnormal liver or renal function (more than twice the normal upper limit of the research institute)
* Uncontrolled diabetes mellitus (>160 mg/dL of fasting blood sugar)
* History of fracture during the previous year
* Uncontrolled hypertension (>160/100 mmHg)
* Uncontrolled thyroid diseases.
* History of serious cerebro-cardiovascular diseases or cancer such as angina or myocardial infarction within 6 months
* History of any central bone fracture within 1 year
* History of medication for psychiatric diseases such as severe depression, schizophrenia, drug intoxication.
* Alcohol abuser
* Allergic reaction to Ishige Okamurae
* Those who participated in other drug clinical trials within 1 month from the screening date.
* Severe gastrointestinal symptoms such as heartburn and indigestion
* Those who are pregnant, lactating, or plan to become pregnant during the clinical trial
* Those who are judged to be unsuitable by the PI for other reasons

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (score) | 8 weeks
  Gastrointestinal Symptom Rating Scale - questionnaire evaluated at baseline and after 8 weeks. It ranges from the minimum of 0 to the maximum of 75. A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
concentration of high-sensitivity C-reactive protein (mg/L) | 8 weeks
  high-sensitivity C-reactive protein (mg/L) measured at baseline and after 8 weeks
concentration of interferon-γ (pg/mL) | 8 weeks
  interferon-γ (pg/mL) measured at baseline and after 8 weeks
concentration of tumor necrosis factor-α (pg/mL) | 8 weeks
  interferon-γ (pg/mL) measured at baseline and after 8 weeks measured at baseline and after 8 weeks
concentration of gastrin (pg/mL) | 8 weeks
  gastrin (pg/mL) measured at baseline and after 8 weeks
concentration of malondialdehyde (mic·mol/L) | 8 weeks
  malondialdehyde (mic·mol/L) measured at baseline and after 8 weeks
concentration of 8-hydroxy-2' -deoxyguanosine (ng/100 mg of protein) | 8 weeks
  8-hydroxy-2' -deoxyguanosine (ng/100 mg of protein) measured at baseline and after 8 weeks
Nepean dyspepsia index-Korean version (score) | 8 weeks
  Nepean dyspepsia index-Korean version - questionnaire evaluated at baseline and after 8 weeks. It ranges from the minimum of 0 to the maximum of 195. A higher score indicates a worse outcome.
Nepean dyspepsia index-Korean version QOL questionnaire (score) | 8 weeks
  Nepean dyspepsia index-Korean version QOL questionnaire evaluated at baseline and after 8 weeks. It ranges from the minimum of 0 to the maximum of 125. A higher score indicates a worse outcome.
Gastrointestinal symptom scale (score) | 8 weeks
  Gastrointestinal symptom scale questionnaire evaluated at baseline and after 8 weeks. It ranges from the minimum of 0 to the maximum of 40. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No